CLINICAL TRIAL: NCT00004059
Title: A Phase I Study of the Cyclin-Dependent Kinase (CDK)/Protein Kinase C (PKC) Inhibitor UCN-01 (NSC 638850) in Combination With 5-Fluorouracil in Patients With Advanced Solid Tumors
Brief Title: Fluorouracil Plus UCN-01 in Treating Patients With Advanced or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-024; CDR0000067256 (Registry Identifier: PDQ (Physician Data Query)); NCI-T99-0037
Record Dates: First submitted 1999-12-10; First posted 2003-05-08 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 7-hydroxystaurosporine; Fluorouracil

INTERVENTIONS:
Drug: 7-hydroxystaurosporine
Drug: fluorouracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. UCN-01 may increase the effectiveness of a chemotherapy drug by making tumor cells more sensitive to the drug.

PURPOSE: Phase I trial to study the effectiveness of fluorouracil plus UCN-01 in treating patients who have advanced or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose, dose limiting toxicity, and toxicity profile of fluorouracil with UCN-01 in patients with advanced or refractory solid tumors.
* Assess the clinical pharmacokinetics of this regimen and correlate with observed toxicities in these patients.
* Obtain preliminary data on the therapeutic activity of this regimen in these patients.

OUTLINE: This is a dose escalation study of fluorouracil.

Patients receive fluorouracil IV over 24 hours on days 1, 8, 15, and 22. Patients receive an initial dose of UCN-01 IV over 72 hours beginning on day 2 during course 1 and then maintenance UCN-01 IV over 36 hours beginning on day 2 during subsequent courses. Treatment repeats every 4 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of fluorouracil until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 6-48 patients will be accrued for this study within approximately 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor that is refractory to standard therapy or for which no standard therapy exists
* Measurable or evaluable disease
* No CNS metastasis or primary CNS malignancy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT and SGPT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No history of coronary artery disease documented by prior myocardial infarction, angiography, or coronary-artery bypass grafting
* No cardiac arrhythmias or congestive heart failure within the past 6 months
* Stable atrial fibrillation on standard treatment allowed at discretion of investigator

Pulmonary:

* DLCO at least 60% of predicted

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study
* No active serious or uncontrolled infection
* HIV negative
* No diabetes
* No other medical condition that would preclude study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered
* Prior fluorouracil allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior mediastinal radiotherapy
* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No concurrent anticonvulsant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States